CLINICAL TRIAL: NCT02063230
Title: An Open-label, Comparative Study to Assess the Pharmacokinetics, Safety and Tolerability of Selumetinib (AZD6244, ARRY-142886) (Hyd-Sulfate) Following Single Oral Dosing to Healthy Subjects and to Subjects With Mild, Moderate, and Severe Hepatic Impairment
Brief Title: To Assess the Pharmacokinetics, Safety and Tolerability of Selumetinib in Patients With Hepatic Impairment and Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D1532C00082
Record Dates: First submitted 2014-02-13; First posted 2014-02-14 (Estimated); Results first posted 2015-11-02 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-06

CONDITIONS: Solid Tumors
Keywords: Phase I, healthy, pharmacokinetic, hepatic impairment
MeSH Terms: interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Selumetinib HV (Experimental): Healthy volunteers (HV)
  Interventions: Drug: Selumetinib 50mg
- Selumetinib mild impairment (Experimental): Mild (Child Pugh A) hepatic impaired patients
  Interventions: Drug: Selumetinib 50mg
- Selumetinib moderate impairment (Experimental): Moderate (Child Pugh B) hepatic impaired patients
  Interventions: Drug: Selumetinib 50mg
- Selumetinib severe impairment (Experimental): Severe (Child Pugh C) hepatic impairment patients
  Interventions: Drug: Selumetinib 25mg

INTERVENTIONS:
Drug: Selumetinib 50mg — HV and hepatic impaired patients with mild and moderat severity will recived selumetinib 50mg orally on day 1
  Arms: Selumetinib HV; Selumetinib mild impairment; Selumetinib moderate impairment
Drug: Selumetinib 25mg — Severe (Child Pugh C) hepatic impaired patients will receive selumetinib 25mg orally on Day 1
  Arms: Selumetinib severe impairment

SUMMARY:
A study to assess the pharmacokinetics, safety and tolerability of Selumetinib (AZD6244, ARRY-142886) in patients with hepatic impairment and healthy subjects.

DETAILED DESCRIPTION:
An open label study to assess the pharmcokinetics, safety and tolerability of a single dose of Selumetinib (AZD6244, ARRY-142886) in patients with hepatic impairment and healthy subjects.

ELIGIBILITY:
Inclusion Criteria for all participants:

1. Subjects will be males or females (non-childbearing potential) aged 18 years or more and with a weight of at least 45 kg and a BMI between 18 and 40 kg/m2 inclusive.

   Inclusion Critera only for hepatic impaired patients:
2. Subjects with stable liver cirrhosis and hepatic impairment for at least 3 months prior to the start of the study.

   Inclusion Criteria only for healthy volunteers:
3. Subjects must be in good health, as determined by a medical history, physical examination, 12-lead ECG, clinical laboratory evaluations, and an ophthalmic examination performed before the administration of the investigational product.

Exclusion Criteria for all participants:

1. Subjects of Japanese or non-Japanese Asian ethnicity
2. Any one parent or grandparent (maternal or paternal) is Japanese or non-Japanese Asian (eg, China, Taiwan, Korea, Philippines, Thailand, Vietnam, and Malaysia). Asian Indians are acceptable.
3. Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of the investigational product
4. Subjects who smoke more than 10 cigarettes or the equivalent in tobacco per day.

   Exclusion criteria for hepatic impaired patients only
5. Undergone liver transplantation. -

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Marbury, MD, Principal Investigator — Orlando Clinical Research Center, 5055 S Orange Avenue, Orlando, Florida, United States.; Ian Smith, MD, Study Director — Astrazeneca, UK
Locations (1):
- Research Site, Orlando, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Mild: Mild (Child Pugh A) hepatic impaired subjects (all subjects received Selumetinib 50 mg)
- Moderate: Moderate (Child Pugh B) hepatic impaired subjects). 6 subjects received Selumetinib 50 mg, 2 received Selumetinib 25mg
- Severe: Severe (Child Pugh C) hepatic impaired subjects. All subjects received Selumetinib 20mg.
- Normal: Healthy volunteers. All volunteers received Selumetinib 50mg.
Period: Overall Study
Arm/Group | Mild | Moderate | Severe | Normal
Started | 8 | 8 | 8 | 8
Received Treatment | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild | Moderate | Severe | Normal | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55 (4) | 57 (5) | 55 (9) | 57 (7) | 56 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 | 3 | 9
  Male | 7 | 5 | 6 | 5 | 23

OUTCOME MEASURES:

1. Primary Outcome: AUC (0 to Infinity) of Total Selumetinib
Time Frame: 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post dose
Population: In the moderate group, 2 patients received Selumetinib 25mg and are not included here but are included in the Dose Normalised AUC outcome measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Mild | Moderate | Severe | Normal
Number analyzed (Participants) | 8 | 6 | 8 | 8
ng*h/mL | 2300 (38.9) | 4300 (45.3) | 1680 (19.9) | 2680 (37.3)

2. Primary Outcome: Cmax of Total Selumetinib
Time Frame: 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post dose
Population: In the moderate group, 2 patients received Selumetinib 25mg and are not included here but are included in the Dose Normalised Cmax outcome measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Mild | Moderate | Severe | Normal
Number analyzed (Participants) | 8 | 6 | 8 | 8
ng/mL | 741 (47) | 1210 (43.2) | 370 (49.8) | 944 (37.0)

3. Primary Outcome: Dose Normalized AUC, Total Selumetinib
Time Frame: 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/mg
Arm/Group | Mild | Moderate | Severe | Normal
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng*h/mL/mg | 45.9 (39.0) | 85.1 (38.3) | 84.3 (20.1) | 53.6 (37.3)

4. Primary Outcome: Dose Normalized Cmax, Total Selumetinib
Time Frame: 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Mild | Moderate | Severe | Normal
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng/mL/mg | 14.8 (47.0) | 23.6 (37.4) | 18.5 (49.9) | 18.9 (37.0)

5. Primary Outcome: Dose Normalized AUC, Unbound Selumetinib
Time Frame: 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/mg
Arm/Group | Mild | Moderate | Severe | Normal
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng*h/mL/mg | 0.127 (41.4) | 0.259 (53.0) | 0.583 (44.9) | 0.184 (30.2)

6. Primary Outcome: Dose Normalized Cmax, Unbound Selumetinib
Time Frame: 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Mild | Moderate | Severe | Normal
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng/mL/mg | 0.0409 (55.4) | 0.0716 (51.0) | 0.128 (73.0) | 0.0647 (32.0)

ADVERSE EVENTS:
Arm/Group | Mild | Moderate | Severe | Normal
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 2/8 | 0/8 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild (N=8) | Moderate (N=8) | Severe (N=8) | Normal (N=8)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head Ache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
In the moderate group, 2 patients received Selumetinib 25mg and are not included in sumaries for AUC and Cmax. Dose normalized parameters are more appropriate for comparisons between groups and are included for all subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No